CLINICAL TRIAL: NCT06874595
Title: Psychobiological Responses Following Exercise and Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20031307
Record Dates: First submitted 2025-02-04; First posted 2025-03-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Psychological
Keywords: Exercise and Brain Stimulation
MeSH Terms: conditions — Motor Activity | interventions — Recombinational DNA Repair; Exercise

STUDY DESIGN:
Intervention Model Description: Repeated measures design; same subjects, same dependent variables across multiple time points, during three conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- High density transcranial direct current stimulation (HD-tDCS) (Experimental): HD-tDCS (High-definition transcranial direct current stimulation) is a novel non-invasive brain stimulation (NIBS) technique based on the principle that when weak intensity electric currents are targeted on specific areas of the scalp, they cause underlying cortical stimulation.
  Interventions: Other: Cycling exercise at 65% of HRR for 20 minutes followed by HD-tDCS (exercise + HD-tDCS); Other: Cycling exercise at 65% of HRR exercise followed by sham HD-tDCS (exercise + sham tDCS); Other: No exercise followed by HD-tDCS (no exercise + HD-tDCS).; Other: State Anxiety Inventory; Other: Visual Analog Scale for Anxiety

INTERVENTIONS:
Other: Cycling exercise at 65% of HRR for 20 minutes followed by HD-tDCS (exercise + HD-tDCS) — Subject will complete a Cycling exercise at 65% of HRR for 20 minutes and then a High-definition transcranial direct current stimulation (HD-tDCS) is a non-invasive brain stimulation technique that uses small electrodes to deliver weak electric currents to the scale. Transcranial direct current stimulation (tDCS) uses weak direct currents of the order of 0.5 mA to 4 mA to modulate cortical activity by exciting or suppressing underlying neurons.
Other: Cycling exercise at 65% of HRR exercise followed by sham HD-tDCS (exercise + sham tDCS) — Subject will complete a Cycling exercise at 65% of HRR for 20 minutes and then a sham High-definition transcranial direct current stimulation (HD-tDCS) is a non-invasive brain stimulation technique that uses small electrodes to deliver weak electric currents to the scale. Transcranial direct current stimulation (tDCS) uses weak direct currents of the order of 0.5 mA to 4 mA to modulate cortical activity by exciting or suppressing underlying neurons.
Other: No exercise followed by HD-tDCS (no exercise + HD-tDCS). — No exercise but a High-definition transcranial direct current stimulation (HD-tDCS) is a non-invasive brain stimulation technique that uses small electrodes to deliver weak electric currents to the scale. Transcranial direct current stimulation (tDCS) uses weak direct currents of the order of 0.5 mA to 4 mA to modulate cortical activity by exciting or suppressing underlying neurons.
Other: State Anxiety Inventory — A widely used psychological assessment tool designed to measure both state and trait anxiety. 40 self-report items rated on a 4-point Likert scale (1 = "Almost Never" to 4 = "Almost Always"). Higher scores indicate higher levels of anxiety. Scores are compared to normative data to determine if they fall within the range of typical or clinical anxiety.
Other: Visual Analog Scale for Anxiety — The Visual Analogue Scale for Anxiety (VASA) is a 100-millimeter line that helps people measure how anxious they feel. The scale has a mark on the left end that indicates "not at all anxious" and a mark on the right end that indicates "very anxious".

SUMMARY:
Anxiety disorders are the most common mental health diagnosis in the US; 19.1% of U.S. adults (23.4% for females and 14.3% for males). In addition, the Global Burden of Disease study (2010) found that anxiety disorders were the sixth leading cause of disability (years of life lived with disability). These debilitating disorders are characterized by excessive worry and fear about everyday situations, and physical symptoms including restlessness, being easily fatigued, difficulty concentrating, irritability, muscle tension, or sleep disturbance. Furthermore, anxiety is linked to other mental disorders including depression and substance abuse; is associated with cardiovascular disease risk factors and a higher rate of cardiovascular disease; and is related to premature mortality. These data have led to the investigation of a breadth of plausible treatments for anxiety, including medications and psychotherapy. However, likely due to the breadth of complex mechanisms involved in the pathophysiology of anxiety disorders and the unfavorable side effects of various medications, a considerable number of individuals do not have a satisfactory response to these treatments. This has led investigators to examine plausible novel interventions to alleviate anxiety and its symptoms.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS), a non-invasive central neuromodulatory technique that is inexpensive and safe, has been utilized to stimulate specific regions of the brain and has demonstrated promising results for alleviating anxiety and depression. (1) evidence supports the administration of anodal stimulation over the left dorsolateral prefrontal cortex (DLPFC) to excite neuronal activity and cathodal stimulation over the right DLPFC to inhibit activity (a bicephalic tDCS montage with 2 mA of stimulation at the left DLPFC) as the most effective tDCS treatment to alleviate anxiety in humans and (2) that "tDCS may be more effective when used in combination with drugs and cognitive behavioral therapies". However, results from studies that have examined the neurophysiological and behavioral effects of tDCS are not consistent. This is likely because the highest cortical current density may not have occurred directly under the target electrode, thus altering the effects of tDCS. High-density tDCS (HD-tDCS) is similar to conventional tDCS utilizing anode and cathode placement on the scalp to produce unidirectional current flow, however, to enhance precision and accuracy, HD-tDCS utilizes smaller electrodes and most often in a "4X1 ring" montage (center anode electrode surrounded by four return cathode electrodes). This HD-tDCS montage delivers a precise current to the intended target site and has been found to be well tolerated and safe for healthy humans. Furthermore, the utilization of HD-tDCS can facilitate the elucidation of mechanisms of action that can provide greater clarity regarding discrepant results in the literature and for considering future advancements in enhancing effective HD-tDCS implementation strategies. HD-tDCS stimulation increases the membrane potential by several millivolts without triggering an action potential.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* aged 18 to 50
* consent and complete a Physical Activity Readiness Questionnaire (PAR-Q)
* be free from any neurological or psychiatric disorder
* not be taking any medication that could affect the central nervous system
* not have any contraindication for HD-tDCS (i.e. not having metal implanted in the head, pacemaker, medical bumps, seizures, lesions on the scalp or head ) or for bioelectrical impedance (i.e., electronic medical implant, such as a pacemaker or implantable cardioverter defibrillator, and limb amputation)
* not be regular users of tobacco products (cigarettes, cigars, chewing tobacco)
* not consume an average of more than ten alcoholic beverages per week

Exclusion Criteria:

* Individuals who do not meet the PAR-Q screening criteria for participation in moderate physical activity will be excluded from participating in this study
* women who are pregnant will be exclude from this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Examine the anxiolytic effects of high density transcranial direct current stimulation (HD-tDCS) "primed" with physical activity (PA) | Completion of 4 visits to research laboratory up to 15 days
  Physical activity prior to HD-tDCS will enhance the anxiolytic effects beyond the benefits of physical activity alone and HD-tDCS alone. Thus, demonstrating a priming effect of PA on the anxiety alleviating electrical pathways that HD-tDCS activates at subthreshold level. Visual Analog Scale for Anxiety (VAS-Anxiety; rating from 0 = "not at all anxious" to 100 = "the most anxious I have ever felt") and three other scales assessing tingling, stiffness and numbness will be administered with a similar VAS

SECONDARY OUTCOMES:
Cerebral hemodynamics assessment | Completion of 4 visits to research laboratory up to 15 days
  Cerebral hemodynamics will be assessed utilizing a Portalite near-infrared spectroscopy (NIRS) device . Changes in cerebral hemodynamics are strongly correlated, both spatially and temporally, with changes in neural activity. The Portalite NIRS system utilizes near-infrared light, which penetrates the skull and brain but is absorbed by hemoglobin (Hb) chromophores in capillary, arteriolar, and venular beds
HRV parameters will be acquired and calculated | Completion of 4 visits to research laboratory up to 15 days
  IHRV parameters will be calculated using the HRV analysis function included in the Biopac AcqKnowledge software. The root mean square of successive differences between normal heartbeats (RMSSD) is obtained by calculating each successive time difference between heartbeats in milliseconds. Then, each of the values is squared and the result is averaged before the square root of the total is obtained. The RMSSD reflects the beat-to-beat variance in HR and is the primary time-domain measure used to estimate the vagally mediated changes reflected in HRV. In addition, low frequency (LF) and high frequency (HF) HRV parameters will be computed in absolute power (ms2). High frequency (HF: 0.15-0.4 Hz) is associated with parasympathetic activity and low frequency (LF: 0.04 - 0.15 Hz) is related to both parasympathetic and sympathetic activity, as it may represent baroreflex-mediated autonomic nervous system (ANS) modulation.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Acevedo, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States